CLINICAL TRIAL: NCT03437720
Title: A 52-week Double-blind, Randomized, Placebo-controlled, Phase 2 Study to Assess the Efficacy and Safety of SAR425899 for the Treatment of Non-alcoholic Steatohepatitis (NASH)
Brief Title: Assessment of the Safety and Effect of SAR425899 Versus Placebo for the Treatment of Non-alcoholic Fatty Liver Disease
Acronym: Restore
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to cancel TRIAL, not related to safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT15067; 2017-002371-26 (EudraCT Number); U1111-1191-5486 (Other: UTN)
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Non-alcoholic Steatohepatitis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — SAR425899

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAR425899 (Low Dose) (Experimental): Once daily dose with weekly dose escalations, if tolerated, until target dose is reached. From week 14 (Day 99) until week 52, no further dose adjustments are planned.
  Interventions: Drug: SAR425899
- SAR425899 (High Dose) (Experimental): Once daily dose with weekly dose escalations, if tolerated, until target dose is reached. From week 14 (Day 99) until week 52, no further dose adjustments are planned.
  Interventions: Drug: SAR425899
- Placebo (Low Dose) (Placebo Comparator): Once daily dose with weekly dose escalations, if tolerated, until target dose is reached. From week 14 (Day 99) until week 52, no further dose adjustments are planned.
  Interventions: Drug: Placebo
- Placebo (High Dose) (Placebo Comparator): Once daily dose with weekly dose escalations, if tolerated, until target dose is reached. From week 14 (Day 99) until week 52, no further dose adjustments are planned.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR425899 — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous injection
  Arms: SAR425899 (High Dose); SAR425899 (Low Dose)
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous injection
  Arms: Placebo (High Dose); Placebo (Low Dose)

SUMMARY:
Primary Objective:

- To evaluate the dose response relationship of SAR425899 compared to placebo on resolution of non-alcoholic steatohepatitis (NASH) with no worsening of fibrosis in diabetic and non-diabetic patients with histopathologically-confirmed NASH.

Secondary Objectives:

* To assess the effect of SAR425899 on overall non-alcoholic fatty liver disease (NAFLD) activity score (NAS), individual components of NAS (steatosis, hepatocyte ballooning, and lobular inflammation), and fibrosis score.
* To assess to the effect of SAR425899 on MRI-PDFF (Magnetic Resonance Imaging-determined Proton Density Fat Fraction) derived parameters (total liver fat, liver volume, and fractional liver fat content).
* To assess the effect of SAR425889 on body weight and waist/hip circumference ratio.
* To assess SAR425899 pharmacokinetics.
* To assess safety and tolerability of SAR425899.

DETAILED DESCRIPTION:
Study duration per participant will be approximately 64 weeks, consisting of up to 8 weeks screening plus 52 weeks treatment and 4 weeks post treatment follow-up.

ELIGIBILITY:
Inclusion criteria :

* Non-diabetic or type 2 diabetes mellitus with confirmed non-alcoholic steatohepatitis.
* Non-alcoholic fatty liver disease (NAFLD) activity score (NAS) >=4 with each of its components >=1.
* Patients without Type 2 diabetes determined by HbA1c (glycated hemoglobin) <6.5% and Fasting Plasma Glucose (FPG) <7.0 mmol/L (<126 mg/dL).
* Stable glycemic control (HbA1c <9.0%) and metabolic disorders managed with diet/exercise and/or stable dose metformin and/or sulphonylureas for at least 3 months prior to screening (type 2 diabetes patients).
* Signed written informed consent form.

Exclusion criteria:

* Diagnosis of type 1 diabetes mellitus.
* Previous insulin use or use of insulin within the last 6 months, except for episode(s) of short-term treatment (<15 consecutive days) due to intercurrent illness.
* Body Mass Index (BMI) <25 kg/m2 or >45.0 kg/m2.
* Current participation in organized diet/weight reduction program or clinical trial of weight control (within the last 3 months prior to screening), or weight loss attempt, plans for major changes in physical activities or significant change in body weight in the 2 months prior to screening (significant change in body weight is defined as >=5% self-reported change within 6 months prior to randomization if a pre-existing liver biopsy sample was collected prior to screening period.
* Current treatment with glucose-lowering agent(s) other than metformin or sulphonylureas, weight loss drugs including orlistat, systemic steroids, methotrexate, amiodarone, or Vitamin E.
* Alcoholism (past or present) and/or average alcohol consumption per week >21 units (210 g) for males, >14 units (140 g) for females within the last 5 years.
* Poorly controlled hypertension (resting systolic blood pressure (SBP) >160 mm Hg and/or resting diastolic blood pressure (DBP) >95 mm Hg) at screening.
* Some liver diseases, pancreatic disease, liver transplantation and types of cancer.
* Pregnant or breast-feeding women.
* Women of childbearing potential (WOCBP) not protected by highly-effective method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Male subjects, whose partners are able to become pregnant, who do not accept to use a condom during sexual intercourse from study inclusion up to 3 months after last dosing; or who are planning to donate sperm from study inclusion up to 3 months after last dosing.
* Patients with coronary, carotid, or peripheral artery revascularization procedures planned during the screening or treatment phases of the protocol.
* Patients with unstable heart conditions.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-23 (Estimated); Primary Completion 2021-08-25 (Estimated); Study Completion 2021-08-25 (Estimated)

PRIMARY OUTCOMES:
Resolution of Non-alcoholic steatohepatitis (NASH) | Week 52
  Percentage of participants with absence of hepatocyte ballooning (NAFLD - non-alcoholic fatty liver disease - activity score, NAS = 0) without worsening of fibrosis score at week 52. -

SECONDARY OUTCOMES:
No hepatocyte ballooning, lobular inflammation score 0 or 1, without worsening of fibrosis | Week 52
  Percentage of participants with absence of hepatocyte ballooning (NAS = 0), lobular inflammation NAS = 0 or 1, without worsening of fibrosis score at week 52.
Change in overall NAFLD activity score (NAS) | Baseline to week 52
  Change from baseline to week 52 in overall NAFLD activity score (NAS).
Change in NAS individual components | Baseline to week 52
  Change from baseline to week 52 in individual components of NAS (steatosis).
Change in NAS individual components | Baseline to week 52
  Change from baseline to week 52 in individual components of NAS (hepatocyte ballooning).
Change in NAS individual components | Baseline to week 52
  Change from baseline to week 52 in individual components of NAS (lobular inflammation).
Change in fibrosis score | Baseline to week 52
  Change from baseline to week 52 in fibrosis score.
Major adverse cardiac events | Baseline to week 52
  Number of patients with major cardiac events
Change in Magnetic Resonance Imaging-determined Proton Density Fat Fraction (MRI-PDFF) | Baseline to week 26 and week 52
  Change from baseline to week 26 and to week 52 in MRI-PDFF-derived total liver fat, liver volume and fractional liver fat content.
Improvement of fibrosis without worsening of hepatocyte ballooning component of NAS | Week 52
  Percentage of participants with improvement of fibrosis by at least 1 stage without worsening of hepatocyte ballooning component of NAS at week 52
Change in body weight | Baseline to week 52
  Change from baseline to week 52 in body weight
Change in waist circumference | Baseline to week 52
  Change from baseline to week 52 in waist circumference
Change in hip circumference | Baseline to week 52
  Change from baseline to week 52 in hip circumference
Change in waist to hip ratio | Baseline to week 52
  Change from baseline to week 52 in waist to hip ratio
Assessment of pharmacokinetic (PK) parameter: AUC0-24 | Week 52
  Area under the concentration-time curve from 0 to 24 hours (AUC0-24)
Assessment of PK parameter: Cmax | Week 52
  Observed maximum plasma concentration after administration (Cmax)
Assessment of PK parameter: Ctrough | Baseline to week 52
  Plasma concentration immediately prior to treatment administration during repeat dosing levels (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org